CLINICAL TRIAL: NCT02777723
Title: Active Controlled, Randomized, Double-blind, Multi-center, Phase 3 Trial to Evaluate the Efficacy and Safety of CKD-350 Eye Drops in Patients With Dry Eye Syndrome
Brief Title: Study to Evaluate the Efficacy and Safety of CKD-350
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 164DES16001
Record Dates: First submitted 2016-05-15; First posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Dry Eye Syndrome
Keywords: Dry Eye Syndrome; Sodium Hyaluronate; CKD-350
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CKD-350 (Experimental): Xenobella
  Interventions: Drug: Xenobella
- Sodium Hyaluronate (Active Comparator): Isotonic 0.3% Sodium Hyaluronate
  Interventions: Drug: Isotonic 0.3% Sodium Hyaluronate

INTERVENTIONS:
Drug: Xenobella — Hypotonic 0.3% Sodium Hyaluronate
  Other Names: Arm A
  Arms: CKD-350
Drug: Isotonic 0.3% Sodium Hyaluronate — Isotonic 0.3% Sodium Hyaluronate
  Other Names: Arm B
  Arms: Sodium Hyaluronate

SUMMARY:
The purpose of this study is to compare the efficacy and safety of CKD-350 in patients with dry eye syndrome

DETAILED DESCRIPTION:
Active controlled, randomized, double-blind, multi-center, phase 3 trial to evaluate the efficacy and safety of CKD-350 eye drops in patients with dry eye syndrome

ELIGIBILITY:
Inclusion Criteria:

1. More than the age of 19 years old
2. Subjects with dry eye symptoms for at least 3 month prior to screening
3. Subjects who have following values 1) ≥ 2 point of corneal staining score 2) ≤ 10 seconds of Tear Break-up Time 3) ≤10mm/5min of Schirmer I Test
4. Subjects who have a visual acuity equal to or better than 0.2 in both eyes
5. Subjects who sign on an informed consent form willingly

Exclusion Criteria:

1. Subjects who have clinically significant ocular surface diseases, abnormal corneal susceptibility and abnormal epiphora
2. Subjects who have medical history following 1) Abnormal eyelids function including abnormality of eyelid or eyelash 2) Ophthalmology operation within 1 year 3) Active ocular infection at present or treatment of allergic eye diseases 4) Herpetic keratopathy, conjunctiva scar from cicatricial keratoconjunctivitis(alkali injuries, stevens-johnson syndrome, ocular cicatricial pemphigoid), pterygium, congenital lacrimal gland absence, neural keratitis, keratoconus
3. Subjects who have received occlusion therapy with lacrimal or punctal plugs within 3 months or have a surgery plan in clinical trial
4. Subjects who wore contact lenses within 3 months or need to wear contact lenses during the study
5. Subjects who take steroidal or immunosuppressive drug within 1 month
6. Over 22mmHg IOP(Intraocular Pressure)
7. Subjects who have malignant tumor within 5 years
8. Subjects with known hypersensitivity to investigational product
9. Women who are nursing, pregnant or planning pregnancy during the study
10. Subjects who have received any other investigational product within 1 month prior to the first dosing
11. Impossible subjects who participate in clinical trial by investigator's decision

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-07 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Changes in Corneal Staining by Oxford scale from Baseline and at Week 4 | Baseline, week 4

SECONDARY OUTCOMES:
Changes in Corneal Staining by Oxford scale from Baseline and at Week 2 | Baseline, week 2
Changes in Tear Break-up Time from Baseline and at Week 2, 4 | Baseline, Week 2, 4
Changes in Schirmer I Test from Baseline and at Week 2, 4 | Baseline, Week 2, 4
Changes in Ocular Surface Disease Index from Baseline and at week 2, 4 | Baseline, week 2, 4

CONTACTS AND LOCATIONS:
Overall Officials: HyoMyung Kim, MD, Study Chair — Korea University Anam Hospital
Locations (14):
- South Korea (14):
  - Chungnam National University Hospital, Daejeon, Chungcheongnam-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Kyungpook National University Hospital, Daegu, Gyeongsangbuk-do
  - Pusan National University Hospital, Pusan, Gyeongsangnam-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Chonnam National University Hospital, Gwangju, Jeollanam-do
  - Asan Medical Center, Seoul, Seoul
  - Gangnam Severance Hospital, Seoul, Seoul
  - Korea University ANAM Hospital, Seoul, Seoul
  - Korea University GURO Hospital, Seoul, Seoul
  - Samsung Medical Center, Seoul, Seoul
  - Seoul National University Hospital, Seoul, Seoul
  - The Catholic University of Korea Seoul ST. MARY'S Hospital, Seoul, Seoul
  - Yonsei University Severance Hospital, Seoul, Seoul

IPD SHARING:
Plan to Share IPD: No